CLINICAL TRIAL: NCT06667817
Title: Exercise From Afar: Progressing At-Risk Rural Adults to Effective Independent Exercise for Dementia Risk Reduction
Brief Title: Exercise From Afar: Progressing At Risk Individuals to Independent Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emporia State University (Other)
Responsible Party: Principal Investigator, Erin Blocker, PI, Emporia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmporiaStateU
Record Dates: First submitted 2024-07-17; First posted 2024-10-31 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Masking Description: Participants will be aware of which study group they are assigned to. Investigators will also be aware of what study group participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): This group will be assigned to the exercise group and will receive the exercise intervention, delivered via the smart phone application.
  Interventions: Behavioral: Exercise
- Control (No Intervention): This group will complete all baseline and follow-up assessments, but receive no intervention. They will serve as the underactive control.

INTERVENTIONS:
Behavioral: Exercise — 16 weeks of exercise training (Exercise Group) will be prescribed via a smart phone application. Results from this group will be compared to results of the sedentary control group.
  Arms: Exercise Group

SUMMARY:
The purpose of this study is to investigate the efficacy of a technology-driven independent exercise program on health outcomes associated with dementia risk among underactive rural adults.

Underactive adults (n=50), ages 40-70 years, from federally designated rural and frontier Kansas counties will be recruited to participate in this study. Specific inclusionary and exclusionary criteria will be used to screen potential participants and determine eligibility. Following recruitment and screening, participants will complete baseline physical fitness and health assessments, supervised by the research team. Following completion of baseline assessments, a personal training/fitness app will be employed to design and deliver exercise programming and track exercise participation, adherence and progression over the course of the study. All prescribed exercise will follow national governing body recommendations and include specific exercises found in previous work to be beneficial for physical health and brain plasticity. The study team will record exercise instruction videos that can be accessed by all participants at any time throughout the study. The particular app used will allow the research team to organize exercise videos into structured training sessions, allowing participants to exercise on their own, at the location of their choice, with ample instruction. The app will also allow participants to record themselves performing various exercises and send them to the research team for analysis of technique and safety. Communication between study personnel and participants will be delivered via the app. Phone calls and/or Zoom sessions will be offered as an alternative if necessary. Our goal is to create a safe, effective means of delivering personalized exercise programming to rural adults that reduces barriers to exercise, improves physical fitness and biomarkers associated with dementia risk and lends itself to exercise adherence in a population that is at an increased risk for cognitive decline. Middle aged adults will be included in the study as they are at an age when successful behavior change is more probable (than older, institutionalized adults); older adults will be included as they are in the high-risk category for dementia. Following the exercise intervention, all baseline assessments will be repeated. Data will be compared to determine the impact of the exercise program on each variable (i.e. dementia risk biomarkers, QOL, physical fitness, etc.).

DETAILED DESCRIPTION:
Following screening, participants will complete baseline physical fitness and health assessments, supervised by the research team. This will require travel by the research team to various rural Kansas locations. The assessments will be those considered reliable, validated 'field tests' and can be easily administered with minimal exercise equipment. Assessments will include a submaximal VO2 field test to assess cardiorespiratory fitness, and an estimated 1 repetition maximum test to assess muscular strength.

Assessments will follow ACSM guidelines for safety and progression for middle aged and older adults.

Blood glucose and cholesterol levels will be measured as well, using a device commonly used in the field (Cholestek LDX ™) This device will assess total blood glucose, cholesterol, LDL, HDL and triglycerides. Additional baseline assessments may include, but are not limited to: a barriers to being active survey (BBAQ) and a perceived stress survey (PSS). All surveys are attached to this application.

Following completion of baseline assessments, participants will be randomized to one of two groups:

1. Exercise (EX); This group will be given structured exercise programming for 16 weeks.
2. Control (CON); This group will serve as the underactive control for this study. At the end of 16 weeks, they will be offered the same 16-week structured exercise program as the exercise group.

Smart Phone Application A personal training/fitness app will be installed on each participant's smart phone or tablet. The application used will be a highly-rated, commonly used fitness app and will be used in this study to design and deliver exercise programming and track exercise participation, adherence and progression over the course of the study. The study team will record exercise instruction videos that can be accessed by all participants at any time throughout the study. The particular app used will allow the research team to organize exercise videos into structured training sessions, allowing participants to exercise on their own, at the location of their choice, with ample instruction and plentiful exercise modification options.

The app will also allow participants to record themselves performing various exercises and send them to the research team for analysis of technique and safety. Communication between study personnel and participants will be delivered via the app. Phone calls and/or Zoom sessions will be offered as an alternative if necessary. During the initial project period (16 weeks), only the EX group will be given access to the structured exercise plan. Exercise Intervention The exercise intervention will consist of 3 evidence-based exercise sessions weekly for a total of 16 weeks. The target goal for all participants will be 75-150 minutes of aerobic exercise and 2-3 strength training sessions weekly. Exercise will be progressive in nature and participants will be encouraged to achieve the target goal for exercise by week 8 of the study and maintain the target goal for weeks 8-16.

All prescribed exercise will follow national governing body recommendations and include specific exercises found in previous work to be beneficial for physical health and brain plasticity. Following the exercise intervention, all baseline assessments will be repeated. Data will be compared to determine the impact of the exercise program on each variable (i.e. dementia risk biomarkers, BBAQ, PSS, and physical fitness.). In order to be included for data analysis, participants must complete 40 of the 48 exercise sessions (i.e. 83% of the sessions)

ELIGIBILITY:
Inclusion Criteria:

* 40 to 70 years of age
* Characterized as underactive by the TAPA
* Able to read and converse in English
* Willing and able to install an application on their smart phone

Exclusion Criteria:

* Myocardial infarction or symptoms of coronary artery disease in the last 2yrs
* Uncontrolled hypertension within the last 6 months
* Cancer in the last 2yrs (except non-metastatic basal or squamous cell carcinoma)
* Significant pain or musculoskeletal disorder that would prohibit participation in an exercise program
* Possible/probably dementia or mild cognitive impairment (MCI) base on adjudication
* Physician concern regarding safety or completion of the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Determine the impact of a technology-driven exercise program on exercise adherence. | 16 weeks per participant enrolled
  Exercise log data will be used to determine exercise adherence. Exercise adherence will be reported as the percentage of total exercise sessions completed over the course of the 16-week exercise study period. Exercise adherence will be tracked and recorded for EX participants only, since CON participants will not complete any exercise during the 16-week study period. The investigators hypothesize that Rural adults will report moderate to high adherence (70-80% total sessions completed) over the course of the study.
Determine the impact of a technology-driven exercise program on barriers to being physical active. | 16 weeks per participant enrolled
  Participants will complete the BBAQ (Barriers to Being Active Quiz) at baseline and following the 16-week exercise study period (following 16 weeks of intervention or control). The results will be compared to determine statistical differences, if any, in barriers to participating in exercise between time points and between groups (EX vs CON). Participants assigned to the exercise group will log their exercise using the smart phone application for the entire 16-week study period. Higher scores on the BBAQ equate to a greater number of barriers to being active. The investigators hypothesize that Rural adults will report fewer barriers to being active (lower BBAQ scores) following 16 weeks of the technology-driven exercise intervention.
Determine the impact of a technology-driven exercise program on exercise self-efficacy. | 16 weeks per participant enrolled
  Participants will complete the Exercise Self-Efficacy Scale at baseline and following the 16-week exercise study period (following 16 weeks of intervention or control). The results will be compared to determine statistical differences, if any, between time points and between groups (EX vs CON). The investigators hypothesize that Rural adults will report higher exercise self-efficacy (higher Self-Efficacy Scale scores) following the intervention (compared to CON participants).
Determine the impact of a technology-driven exercise program on cholesterol and fasting blood glucose. | 16 weeks per participant enrolled
  Fasting blood glucose and cholesterol are measured simultaneously using a Cholestek device. This measure will be completed by all participants at baseline, and again at follow-up (following 16 weeks of intervention or control). The investigators hypothesize that participants in the EX group (exercise intervention) will see greater improvements in total cholesterol, fasting blood glucose and LDL following the intervention, compared to the CON group. The investigators expect that participants with higher exercise adherence will see the greatest improvements in these biomarkers associated with reduced dementia risk.
Determine the impact of a technology-driven exercise program on cardiorespiratory fitness. | 16 weeks per participant enrolled
  Participants will also complete a common cardiorespiratory field test at baseline and again at follow-up (after 16 weeks of intervention or control). The investigators hypothesize that cardiorespiratory fitness scores will improve for EX participants following the 16-week intervention and that the post-intervention cardiorespiratory field test scores will be significantly better than those of the CON group.
Determine the impact of a technology-driven exercise program on muscular fitness. | 16 weeks per participant enrolled
  Participants will complete an repetition maximum muscular fitness test at baseline and again at follow-up (after 16 weeks of intervention or control). The investigators hypothesize that muscular fitness will improve for EX participants following the 16-week intervention and that the post-intervention muscular fitness results will be significantly better than those of the CON group.

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Blocker, PhD, Principal Investigator — Emporia State University
Locations (1):
- Emporia State University, Emporia, Kansas, United States

DOCUMENTS (3):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT06667817/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT06667817/SAP_001.pdf
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT06667817/ICF_002.pdf